CLINICAL TRIAL: NCT02162251
Title: Post-marketing Surveillance of Donepezil Hydrochloride Investigation of the Safety and Effectiveness of Combination Therapy of Donepezil Hydrochloride and Memantine Hydrochloride in Patients With Alzheimer's Disease
Status: Completed | Type: Observational
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Other Study IDs: ART07T
Record Dates: First submitted 2014-06-10; First posted 2014-06-12 (Estimated); Last update posted 2018-09-07 (Actual); Status verified 2016-12

CONDITIONS: Alzheimer's Desease
Keywords: Alzheimer's Disease; donepezil hydrochloride
MeSH Terms: conditions — Alzheimer Disease | interventions — Donepezil

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- E2020
  Interventions: Drug: Donepezil Hydrochloride

INTERVENTIONS:
Drug: Donepezil Hydrochloride — Initial dose of 3 mg orally once daily. After 1-2 weeks, dosage increased to 5 mg orally once daily. After 4 or more weeks, dosage increased to 10 mg orally once daily for patients with severe dementia of Alzheimer's type. Dose reduced appropriately according to patient's symptoms.
  Other Names: Aricept

SUMMARY:
To investigate the safety and effectiveness about administration of both donepezil hydrochloride and menatine hydrochloride in patients with Alzheimer's Disease in clinical practice.

ELIGIBILITY:
Inclusion criteria:

Patients diagnosed with Alzheimer's Disease who are to be administered both donepezil hydrochloride and memantine hydrochloride in clinical practice.

Exclusion criteria:

Patients with a history of hypersensitivity to any ingredients of Aricept or piperidine derivatives.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Alzheimer's Disease
Sampling Method: Non-Probability Sample
Enrollment: 3482 (Actual)
Dates: Start 2013-06-01 (Actual); Primary Completion 2015-05-01 (Actual); Study Completion 2016-04-15 (Actual)

PRIMARY OUTCOMES:
Investigations on adverse events and adverse drug reactions | Up to 12 months

SECONDARY OUTCOMES:
Severity of dementia based on the Functional Assessment Staging Test (FAST) | Baseline, Month 3, Month 6, and Month 12
  FAST is a seven stage system based on level of functioning and daily activities. It focuses more on an individual's level of functioning and activities of daily living versus cognitive decline
Change From Baseline in the Mini-Mental State Examination (MMSE) Score | Baseline and Month 12
  The MMSE is a brief 30-point questionnaire test that is used for the assessment of dementia patients' cognitive impairment. Evaluation of points are as follows: 24 to 30 = no cognitive impairment, 18 to 23 = mild cognitive impairment, 0 to 17 = severe cognitive impairment. Lower scores indicate worsening.

CONTACTS AND LOCATIONS:
Locations (1):
- Multiple Locations, Japan

REFERENCES:
- [Result] Geriatric Medicine 55(1): 87-100, 2017.
- [Result] Geriatric Medicine 55(11): 1251-1264, 2017.